CLINICAL TRIAL: NCT06882603
Title: Comparison of the Efficacy of Corticosteroid Injection and Saline Nerve Hydrodissection on Electrophysiological Study, Pain, Function and Sonographic Findings in the Treatment of Carpal Tunnel Syndrome: A Randomized Controlled Trial
Brief Title: Efficacy of Corticosteroid Injection and Nerve Hydrodissection in Carpal Tunnel Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Basak Cigdem Karacay, associate professor, Kirsehir Ahi Evran Universitesi
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024/470
Record Dates: First submitted 2025-03-11; First posted 2025-03-18 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Carpal Tunnel Syndrome (CTS)
Keywords: steroid injection; nerve hydrodissection
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Steroids; Exercise

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigator and outcomes assessor are different people.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Steroid injection (Experimental): The Group 1 under steroid injection + tendon and median nerve gliding exercise
  Interventions: Other: Steroid injection; Other: Exercise
- Hydrodissection (Experimental): The Group 2 under hydrodissection + tendon and median nerve gliding exercise
  Interventions: Other: hydrodissection; Other: Exercise
- Exercise (Other): Group 3 under tendon and median nerve gliding exercise
  Interventions: Other: Exercise

INTERVENTIONS:
Other: hydrodissection — 5 ml of 0.9% isotonic sodium chloride solution will be applied to the intracarpal area median nerve area once with the USG probe.
  Arms: Hydrodissection
Other: Steroid injection — 1 ml of 3mg/ml betamethasone sodium phosphate or 3mg/ml betamethasone acetate solution will be applied with the USG probe.
  Arms: Steroid injection
Other: Exercise — Performed with 6 different consecutive positions of the hand and wrist. 1- Wrist in neutral position, fingers and thumb in flexion 2- Wrist in neutral position, fingers and thumb in extension 3- Wrist and fingers in extension, thumb in neutral position 4- Wrist, fingers and thumb in extension 5- Forearm in supination, wrist and fingers in extension 6- Forearm in supination, wrist and fingers in extension, gentle stretching is applied to the thumb with the hand. Tendon gliding exercises: Performed to ensure isolated mobility of the flexor digitorum superficialis and profundus muscles in the canal. Tendon gliding exercises are performed in 5 different consecutive positions, respectively. 1- Fingers straight 2- Fingers in hook position 3- Fingers in fist position 4- Fingers in table shape position 5- Fingers in straight fist. The exercises will be asked to be done 10 times, once a day, every day for 3 weeks.

SUMMARY:
The subject of the study is to use current treatment methods in patients with nerve compression in the wrist and compare their effects. The purpose of the study is to determine the most appropriate method by comparing the benefits of cortisone and serum injection in addition to exercise therapy in volunteers like you who have nerve compression in the wrist and have pain and numbness.

DETAILED DESCRIPTION:
Carpal tunnel syndrome (CTS) was first described by Paget in 1854, and detailed information and surgical techniques regarding its clinical course were provided by Phalen. Carpal tunnel syndrome (CTS) is a clinical picture consisting of symptoms resulting from compression of the median nerve within the carpal tunnel at the wrist level, and is the most common focal entrapment neuropathy. Although it is due to idiopathic and secondary causes, the pathophysiology of CTS is not fully understood. It is 3 times more common in women than in men. The fact that CTS occurs more frequently in the dominant hand supports the important role of hand activity in the development of the disease. Since the sensory branches of the median nerve innervate the first three fingers and half of the 4th finger, CTS patients typically complain of burning, pins and needles, tingling and numbness in these fingers. In some cases, the pain may not correspond to the normal sensory area of the median nerve in the hand. CTS is easily diagnosed by history and physical examination. Imaging and electrodiagnostic studies help confirm the diagnosis. Treatment varies according to the degree of CTS. Different conservative treatment methods are used in the treatment of mild and moderate CTS. The most commonly used methods are splint, local corticosteroid injection (LCE) and conventional treatment agents (TENS, hotpack, ultrasound). Local corticosteroid injection is an injection method with proven efficacy, applied in clinical practice and included in the guidelines. Another method that has become popular recently is hydrodissection of the median nerve. Isotonic sodium chloride solution is injected in the hydrodissection method. It does not contain drugs. Hydrodissection is a minimally invasive procedure that involves injecting fluid into anatomical spaces to facilitate dissection and reduce adhesion during surgery. Smith et al. described lidocaine and corticosteroid injection under ultrasound guidance in patients with CTS and proposed the concept of nerve hydrodissection. The therapeutic effect of nerve hydrodissection is based on the theory that it can separate the nerve from the surrounding soft tissue and reduce the risk of chronic compression injury. The hydrodissection method does not cause side effects related to blood sugar regulation in patients with comorbidities such as diabetes mellitus. Injections under USG guidance both increase the reliability of the injection and are targeted. In this study, all injection procedures will be performed under USG guidance in our clinic.

USG-guided corticosteroid injection is already a procedure applied in the treatment of patients with carpal tunnel syndrome in our clinic. In hydrodissection, the same procedure will be performed under USG guidance and isotonic sodium chloride solution will be used instead of corticosteroid.

The aim of this study is to compare the effectiveness of median nerve hydrodissection with 0.9% isotonic sodium chloride and local corticosteroid injection on electrophysiological studies, pain, function and sonographic findings and to investigate whether it is superior to the control group.

Female and male patients between the ages of 18-65 who apply to Kırşehir Ahi Evran University Hospital PMR outpatient clinic and meet the inclusion criteria will be included in the study. In the prospective randomized controlled single-blind planned study, evaluations will be made at week 0 before treatment, week 3 at the end of treatment and week 12. The estimated number of volunteers expected to participate in the study was determined according to power analysis. The sensory nerve and Tm velocity score, which was the primary outcome measure in the study conducted by Şahin et al. in carpal tunnel syndrome, was taken as reference. The disease will be diagnosed with clinical, physical examination and enmg studies, and no additional techniques will be requested. The patients will be randomly divided into 3 groups. They will be selected by simple random sampling using the closed envelope method and will then be divided into Group 1 (steroid injection + tendon and median nerve gliding exercise), Group 2 (hydrodissection + tendon and median nerve gliding exercise) and Group 3 (tendon and median nerve gliding exercise). The patient will be evaluated with Bostan Carpal Tunnel Syndrome Questionnaire (BCSQT) before treatment, at the end of treatment, in the 3rd and 12th weeks, DN-4 Neuropathic Pain Questionnaire, EMG median sensory nerve conduction velocity and median nerve distal motor latency data, and USG will be used to examine the cross-sectional area of the median nerve at the scaphoid-pisiform bone level.

In this study, three different treatment methods will be grouped in three different ways.

ELIGIBILITY:
Inclusion Criteria:

1. Female and male patients aged 18-65 who applied to Ahi Evran University Physical Medicine and Rehabilitation Polyclinic and diagnosed with carpal tunnel syndrome through clinical and EMG
2. Patients who can understand the information form correctly and are cooperative
3. Patients who consented to participate in the study according to the informed consent form

Exclusion Criteria:

1. Cervical radiculopathy
2. Polyneuropathy
3. Brachial plexopathy
4. Systemic corticosteroid use
5. History of fracture and trauma in the forearm and wrist on the treated side 6- Inflammatory rheumatic disease

7- Pregnant and breastfeeding patients 8- Systemic diseases such as renal failure, peptic ulcer, diabetes, hypothyroidism, coagulation disorders 9- Patients who have undergone carpal tunnel syndrome surgery 10- Thoracic outlet syndrome 11- Thenar atrophy, severe carpal tunnel syndrome 12- Patient is unwilling or states that they cannot participate for any reason

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-10-14 (Actual); Primary Completion 2026-02-05 (Estimated); Study Completion 2026-05-05 (Estimated)

PRIMARY OUTCOMES:
Electrophysiological Study | 0 day
  All patients will undergo electroneurophysiological examination at the EMG laboratory of the Neurology Department of Kırşehir Ahi Evran University Education and Research Hospital before treatment and at 12 weeks after treatment.Median sensory nerve action potential amplitude, Compound muscle action potential amplitude, Median sensory distal latency, Median motor distal latency, Median sensory nerve conduction velocity, was evaluated by EMG.
Electrophysiological Study | 12th week
  All patients will undergo electroneurophysiological examination at the EMG laboratory of the Neurology Department of Kırşehir Ahi Evran University Education and Research Hospital before treatment and at 12 weeks after treatment.Median sensory nerve action potential amplitude, Compound muscle action potential amplitude, Median sensory distal latency, Median motor distal latency, Median sensory nerve conduction velocity, was evaluated by EMG.

SECONDARY OUTCOMES:
Measurement of the median nerve cross-sectional area with USG | 0 day
  The use of ultrasonography in the evaluation of CTS is increasing. To measure the median nerve cross-sectional area, the nerve is determined with a continuous line along the hyperechoic border, and the cross-sectional area of the circled area will be calculated with USG.
Measurement of the median nerve cross-sectional area with USG | 4th week
  The use of ultrasonography in the evaluation of CTS is increasing. To measure the median nerve cross-sectional area, the nerve is determined with a continuous line along the hyperechoic border, and the cross-sectional area of the circled area will be calculated with USG.
Measurement of the median nerve cross-sectional area with USG | 12th week
  The use of ultrasonography in the evaluation of CTS is increasing. To measure the median nerve cross-sectional area, the nerve is determined with a continuous line along the hyperechoic border, and the cross-sectional area of the circled area will be calculated with USG.
Boston Carpal Tunnel Questionnaire | 0 day
  The Boston Carpal Tunnel Syndrome Questionnaire, which has been validated and reliable in Turkish (10), has been proposed for clinical standardization of carpal tunnel syndrome patients. The questionnaire consists of nineteen questions and the answers are evaluated with a minimum of one and a maximum of five points. The lowest score is 5 and the highest score is 95. A high average score indicates that the patient's complaints are severe or that their functional capacity is inadequate.
Boston Carpal Tunnel Questionnaire | 4th week
  The Boston Carpal Tunnel Syndrome Questionnaire, which has been validated and reliable in Turkish (10), has been proposed for clinical standardization of carpal tunnel syndrome patients. The questionnaire consists of nineteen questions and the answers are evaluated with a minimum of one and a maximum of five points. The lowest score is 5 and the highest score is 95. A high average score indicates that the patient's complaints are severe or that their functional capacity is inadequate.
Boston Carpal Tunnel Questionnaire | 12th week
  The Boston Carpal Tunnel Syndrome Questionnaire, which has been validated and reliable in Turkish (10), has been proposed for clinical standardization of carpal tunnel syndrome patients. The questionnaire consists of nineteen questions and the answers are evaluated with a minimum of one and a maximum of five points. The lowest score is 5 and the highest score is 95. A high average score indicates that the patient's complaints are severe or that their functional capacity is inadequate.
DN4 Neuropathic Pain Questionnaire | 0 day
  It is an easy-to-use and score tool developed in France. It consists of 4 items, the first two are about the characteristics of the pain and the last two items are about sensory examination findings. A total score of 4 out of 10 indicates neuropathic pain. DN4 has been shown to have 83% sensitivity and 90% specificity. Validity and reliability of the Turkish version were performed by Çelik et al.
DN4 Neuropathic Pain Questionnaire | 4th week
  It is an easy-to-use and score tool developed in France. It consists of 4 items, the first two are about the characteristics of the pain and the last two items are about sensory examination findings. A total score of 4 out of 10 indicates neuropathic pain. DN4 has been shown to have 83% sensitivity and 90% specificity. Validity and reliability of the Turkish version were performed by Çelik et al.
DN4 Neuropathic Pain Questionnaire | 12th week
  It is an easy-to-use and score tool developed in France. It consists of 4 items, the first two are about the characteristics of the pain and the last two items are about sensory examination findings. A total score of 4 out of 10 indicates neuropathic pain. DN4 has been shown to have 83% sensitivity and 90% specificity. Validity and reliability of the Turkish version were performed by Çelik et al.

CONTACTS AND LOCATIONS:
Overall Officials: Basak Cigdem Karacay, Assoc. Prof, Principal Investigator — Kirsehir Ahi Evran Universitesi
Locations (2):
- Turkey (Türkiye) (2):
  - Ahi Evran University, Kırşehir, City Centre
  - Ahi Evran University, Kırşehir

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sahin MA, Cigdem-Karacay B, Konar NM, Tuncay F. Comparison of the Effectiveness of 2 Different Kinesio Taping Techniques Added to Exercises in the Treatment of Carpal Tunnel Syndrome: Randomized Controlled Trial, Double-Blind, Parallel Groups. Arch Phys Med Rehabil. 2024 Sep;105(9):1657-1665. doi: 10.1016/j.apmr.2024.05.023. Epub 2024 Jun 6. PMID 38851555
- [Background] Wu YT, Chen SR, Li TY, Ho TY, Shen YP, Tsai CK, Chen LC. Nerve hydrodissection for carpal tunnel syndrome: A prospective, randomized, double-blind, controlled trial. Muscle Nerve. 2019 Feb;59(2):174-180. doi: 10.1002/mus.26358. Epub 2018 Dec 4. PMID 30339737
- [Background] Wipperman J, Goerl K. Carpal Tunnel Syndrome: Diagnosis and Management. Am Fam Physician. 2016 Dec 15;94(12):993-999. PMID 28075090